CLINICAL TRIAL: NCT05970536
Title: The Effect of Two Different Contemporary Chelating Agents on Vital Pulp Therapy in Mature Permanent Teeth With Irreversible Pulpitis Using Bioceramic Material
Brief Title: Vital Pulp Therapy of Mature Permanent Teeth With Irreversible Pulpitis Using Bioceramic Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Mona Rizk Abo El Wafa Ahmed, principal investigator, Sinai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 341122
Record Dates: First submitted 2023-07-08; First posted 2023-08-01 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-07

CONDITIONS: Vital Pulp Therapy

STUDY DESIGN:
Intervention Model Description: Parallel double blinded.
Who Masked: Participant, Outcomes Assessor
Masking Description: double ( participant, outcome assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apple vinegar group (Experimental): After hemostasis of the exposed pulp is achieved, Apple vinegar will be used for dentin conditioning for 5 mins then 1-2 mm thickness of MTA placed on the exposed pulp chamber.
  Interventions: Other: Apple vinegar or EDTA 17%
- EDTA 17% group (Active Comparator): After hemostasis of the exposed pulp is achieved, EDTA 17 % will be used for dentin conditioning then 1-2 mm thickness of MTA placed on the exposed pulp chamber.
  Interventions: Other: Apple vinegar or EDTA 17%

INTERVENTIONS:
Other: Apple vinegar or EDTA 17% — Application of each chelating agent for 5 minutes for dentin conditioning followed by placement of MTA on the pulp chamber.

SUMMARY:
This clinical trial is designed to study and compare the effect of two different types of chelating agents on the vital pulp therapy of mature permanent teeth with irreversible pulpitis using bioceramic material.

DETAILED DESCRIPTION:
1. The vital pulps exposed by caries process is treated by complete caries removal followed by full pulpotomy.
2. After hemostasis, application of apple vinegar and EDTA 17% will be used followed by MTA application. finally teeth will be restored with resin composite restoration.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one tooth with carious pulp exposure and irreversible pulpitis.
* Cooperative behavior with no medical problem.
* Absence of tooth mobility , tenderness on percussion.
* History of pain with cold and sweets.
* Radiographically, no internal or external resorption, no periapical or furcation radiolucency and no widening of the periodontal membrane space.

Exclusion Criteria:

* Teeth with pulp necrosis.
* Presence of sinus tract.
* Teeth with open apices.
* Pregnant women.
* History of intolerance of non- steroidal anti inflammatory drugs.
* Tenderness to palpation of adjacent soft tissues

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Success rate of vital pulp therapy of mature permanent teeth with irreversible pulpitis using bioceramic material. | one year
  1. Through post operative pain assessment using Visual analogue scale (0-3) scores as 0 represents no pain, 1= mild pain, 2= moderate pain and 3= sever pain. VAS scores marked at intervals of 2,6,24,48 and 72 hours.
  2. Clinical success criteria:
  Clinical parameters indicating successful treatment include the following criteria:
  * Absence of pain except for the first 24 hours.
  * Normal soft tissue around the tooth ( no swelling, no sinus tract).
The Pulp vitality | one year
  Pulp vitality will be assessed through pulpal response to thermal and electrical pulp tests. at 3,6,12 months

SECONDARY OUTCOMES:
Radiographic success | one year
  Using digital periapical radiograph at 3,6,12 months. Radiographic success criteria include:
  * No periapical pathosis.
  * No radicular resorption defects.

CONTACTS AND LOCATIONS:
Overall Officials: Mona R Abo El Wafa Ahmed, PhD, Principal Investigator — Faculty of Dentistry, Sinai University.
Locations (1):
- Mona Rizk Abo El Wafa Ahmed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2 years

REFERENCES:
- [Derived] Sobh YTM, Ahmed MRA. The effect of two different contemporary chelating agents on vital pulp therapy in mature permanent teeth with irreversible pulpitis using bioceramic material: randomized clinical trial. BMC Oral Health. 2024 Aug 8;24(1):918. doi: 10.1186/s12903-024-04627-6. PMID 39118082